CLINICAL TRIAL: NCT00266864
Title: Testosterone Replacement Therapy in Chronic Spinal Cord Injury
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Kessler Institute for Rehabilitation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2648-C
Record Dates: First submitted 2005-12-15; First posted 2005-12-19 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-09

CONDITIONS: Spinal Cord Injury; Hypogonadism
Keywords: Spinal Cord Injury; Testosterone Replacement Therapy; Dual Energy X ray Absorptiometry; Lean Tissue Mass
MeSH Terms: conditions — Spinal Cord Injuries; Hypogonadism | interventions — Testosterone; Transdermal Patch; Testosterone Propionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone Replacement Therapy (Experimental): Subjects with Low Testosterone (Hypogonadal) Receive Testosterone Transdermal System (Androderm 5 mg patch)
  Interventions: Drug: Testosterone Transdermal System (Androderm 5 mg patch)
- No Intervention (No Intervention): Subjects with normal testosterone levels (eugonadal) participated in identical outcome measurements at parallel time points.

INTERVENTIONS:
Drug: Testosterone Transdermal System (Androderm 5 mg patch) — Testosterone Transdermal System (Androderm 5 mg patch)
  Other Names: Androgel (Testim) and Underarm Testosterone (Axiron)
  Arms: Testosterone Replacement Therapy

SUMMARY:
It has long been recognized that co-morbidity associated with multiple metabolic syndrome, such as adverse body composition, insulin resistance and autonomic nervous system impairment, may lead to significant increase in cardiovascular morbidity and mortality. It is unclear whether the co-morbidity evident in this population are due directly to their immobility or are the result of unfavorable changes in their underlying hormonal milieu. The purpose of this study is to determine the effect of testosterone replacement therapy in hypogonadal males on:

body composition, i.e. lean tissue and fat mass, glucose tolerance, resting energy expenditure, autonomic-cardiovascular integrity, muscular strength, psychological assessment

DETAILED DESCRIPTION:
This study is 24 months in duration. Men who have consented to pre-screening serum testosterone draw and are found to have total testosterone levels averaging ≤ 11.3 nmol/l will start testosterone replacement therapy after a 6-month baseline period. Once treatment begins subjects will place a testosterone replacement patch (5 or 10 mg/day) on various sites of the body daily. Subjects will visit the lab after 2,6, 12, and 18 months of therapy for testing; however they will stop taking the patch at the 12 month visit. If needed, a steroid cream will be provided to the subjects should any skin irritations occur. If the patch causes persistent skin irritations, despite use of the steroid cream, then a testosterone gel may be used. Detailed instructions and precautions using the gel are outlined in the consent form and will be reviewed with the subject.

Those men who have consented to pre-screening serum testosterone and are found to have normal levels of total testosterone (testosterone total ≥ 11.4 nmol/l) are eligible to participate as a control subject for the full 24-month period of the study. These subjects visit the lab at baseline (BL), 12 and 24 months for the same testing as those in the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Males 18-49 years of age
* Chronic spinal cord injury
* Normal prostate specific antigen levels and digital rectal exam
* No known cardiovascular disease
* Subjects with total testosterone > 4 ng/ml
* Subjects with total testosterone > 4 ng/ml

Exclusion Criteria:

* Females
* Known coronary heart and/or artery disease, diabetes mellitus
* Previous or current cancer
* Current or previous anabolic steroid use
* Acute inter-current illness
* Abnormal liver function test (>1.5 times normal values) at baseline
* Prostate specific antigen above normal
* Abnormal digital rectal exam at baseline suggestive of malignancy
* Current alcohol or drug abuse
* Significant psychological disorders

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2003-08; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Bauman, MD, Principal Investigator — VA Medical Center, Bronx
Locations (2):
- United States (2):
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - James J. Peters VA Medical Center, The Bronx, New York

REFERENCES:
- [Result] Bauman WA, Cirnigliaro CM, La Fountaine MF, Jensen AM, Wecht JM, Kirshblum SC, Spungen AM. A small-scale clinical trial to determine the safety and efficacy of testosterone replacement therapy in hypogonadal men with spinal cord injury. Horm Metab Res. 2011 Jul;43(8):574-9. doi: 10.1055/s-0031-1280797. Epub 2011 Jun 29. PMID 21717386
- [Result] La Fountaine MF, Wecht JM, Cirnigliaro CM, Kirshblum SC, Spungen AM, Bauman WA. QT/RR coherence is associated with testosterone levels in men with chronic spinal cord injury. Neuroendocrinology. 2011;93(3):174-80. doi: 10.1159/000323773. Epub 2011 Jan 21. PMID 21252493
- [Result] La Fountaine MF, Wecht JM, Cirnigliaro CM, Kirshblum SC, Spungen AM, Bauman WA. Testosterone replacement therapy improves QTaVI in hypogonadal men with spinal cord injury. Neuroendocrinology. 2013;97(4):341-6. doi: 10.1159/000347070. Epub 2013 May 9. PMID 23343764
- [Derived] Bauman WA, La Fountaine MF, Cirnigliaro CM, Kirshblum SC, Spungen AM. Lean tissue mass and energy expenditure are retained in hypogonadal men with spinal cord injury after discontinuation of testosterone replacement therapy. J Spinal Cord Med. 2015 Jan;38(1):38-47. doi: 10.1179/2045772314Y.0000000206. Epub 2014 Jun 26. PMID 24968251
- See also: Click here for more information about this study: Testosterone Replacement Therapy in Chronic Spinal Cord Injury — http://www.unitedspinal.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Testosterone Replacement Therapy: Treatment group: Testosterone Replacement Therapy Patch 5 or 10mg daily (Androderm, Watson Pharma Inc.) for 12 months, with the dose adjusted to raise the serum testosterone concentration to within the normal range.
- No Intervention: Control group: subjects in this group will receive no intervention, but will have the same outcome measures as arm 1 completed at the baseline, 12, and 24 month time points.
Period: Overall Study
Arm/Group | Testosterone Replacement Therapy | No Intervention
Started | 18 | 13
Completed | 13 | 11
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone Replacement Therapy | No Intervention | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 24
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants] — Hypogonadal (Testosterone Replacement Therapy group, total testosterone < 4 ng/ml) and Eugonadal (No Intervention group total testosterone > 4 ng/ml) subjects
  participants
    Male | 13 | 11 | 24
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24
Dual energy x-ray absorptiometry (DXA) for lean tissue mass [Mean (Standard Deviation); unit: kilograms] — Body composition measurements for measures of total body lean tissue mass (LTM) were assessed by dual energy X-ray absorptiometry (DXA; General Electric LUNAR Prodigy Advance, software version 11.4 and 12.2, Madison, WI). In accordance with International Society for Clinical Densitometry guidelines, total body scans were repeated on 30 spinal cord injury subjects by the "on-and-off -the-table" method (i. e., subjects were repositioned between scans) and our precision error was equal to 1.2 % for LTM.
  kilograms | 49.6 (7.6) | 51.9 (8.1) | 50.8 (7.8)
Resting Energy Expenditure [Mean (Standard Deviation); unit: kcal/day] — Resting Energy Expenditure was obtained by the measurement of exhaled air from fractions of mixed expired oxygen and carbon dioxide by a process known as indirect calorimetry. Data was collected under steady state conditions and was adjusted to account for differences in total body lean tissue mass. Participants arrived at the laboratory for testing between the hours of 8:00 and 10:00 in the morning, following a 12 hour fast, with a minimum of 24 hours free from any type of exercise.
  kcal/day | 1328 (262) | 1319 (112) | 1324 (197)

OUTCOME MEASURES:

1. Primary Outcome: Dual Energy X-ray Absorptiometry (DXA) Assessment of Lean Tissue Mass (LTM)
Description: Dual energy X-ray absorptiometry assessment of lean tissue mass (LTM) at 12 months. Total body scans were performed and the energy level used for each total body scan was based on subject thickness (e. g., thin, standard, or thick). To analyze the results of each total body scan, proprietary software algorithms were used to segment the body into trunk, pelvis, and upper and lower extremities using the standard regions of interest. In accordance with International Society for Clinical Densitometry guidelines, total body scans were repeated on 30 spinal cord injury subjects by the "on-and-off -the-table" method (i. e., subjects were repositioned between scans) and our precision error was equal to 1.2 % for LTM.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Testosterone Replacement Therapy | No Intervention
Number analyzed (Participants) | 13 | 11
kilograms | 53.1 (6.9) | 50.5 (6.3)
Statistical Analysis 1: Comparison: Testosterone Replacement Therapy vs No Intervention; Separate 2 factor (group: treatment, control) analysis of variance (ANOVA) with repeated measures on visit (baseline, month 12) were performed to identify changes in lean tissue mass across time. To further characterize significant main and interaction effects, post-hoc paired t -tests were performed within group; Test type: Superiority or Other; p < 0.01, ANOVA — One sample t -tests were performed on the percent change from baseline to month 12 [(month 12- baseline)/baseline*100] for comparison to the null hypothesis. An a priori level of significance was set at p ≤ 0.05; Mean Difference (Final Values) = 3.4, Standard Deviation 2.7

2. Secondary Outcome: Resting Energy Expenditure
Description: Resting Energy Expenditure was obtained by the measurement of exhaled air from fractions of mixed expired oxygen and carbon dioxide by a process known as indirect calorimetry. Data was collected under steady state conditions. Participants arrived at the laboratory for testing between the hours of 8:00 and 10:00 in the morning, following a 12-h fast, with a minimum of 24 h free from any type of exercise.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kcal/day
Groups:
- Testosterone Replacement Therapy: Testosterone Replacement Therapy Patch 5 or 10 mg daily
Arm/Group | Testosterone Replacement Therapy | No Intervention
Number analyzed (Participants) | 13 | 11
kcal/day | 1440 (262) | 1339 (128)
Statistical Analysis 1: Comparison: Testosterone Replacement Therapy vs No Intervention; Separate 2 factor (group: treatment, control) analysis of variance (ANOVA) with repeated measures on visit (baseline, month 12) were performed to identify changes in resting energy expenditure across time. To further characterize significant main and interaction effects, post-hoc paired t -tests were performed within group; Test type: Superiority or Other; p = 0.051, ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 101, Standard Deviation 103

ADVERSE EVENTS:
Time Frame: Adverse events from this study were collected over a 12-month period
Groups:
- Testosterone Replacement Therapy: A prospective, open-label, controlled drug intervention trial was performed in healthy hypogonadal and eugonadal outpatient men with chronic spinal cord injury (Treatment: serum testosterone concentration <4.0 mg/dL and Control: serum testosterone concentration ≥4.0 mg/dL). Treatment subjects received a transdermal testosterone patch (5 or 10 mg; Androderm, Watson Pharma Inc.) daily for 12 months, with the dose adjusted to raise the serum testosterone concentration to within the normal range. Only outcome measures were assessed for the no intervention arm; no adverse events were collected.
Arm/Group | Testosterone Replacement Therapy
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 11/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Replacement Therapy (N=18)
Urinary tract infection (Renal and urinary disorders) | 1 (1) — Autonomic dysreflexia due to urinary tract infection followed by hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Replacement Therapy (N=18)
Skin irritation (Skin and subcutaneous tissue disorders) | 11 (11) — Minor skin irritation at patch site definitely related to testosterone replacement therapy
Acne (Skin and subcutaneous tissue disorders) | 1 (1) — minor body acne probably related to testosterone replacement therapy
Edema (Blood and lymphatic system disorders) | 4 (4) — Increase in lower extremity edema possibly related to testosterone replacement therapy
Elevated hemoglobin and hematocrit (Blood and lymphatic system disorders) | 1 (1) — Slight elevation of hemoglobin and hematocrit levels from testosterone replacement therapy
Liver function enzymes (Hepatobiliary disorders) | 1 (1) — Elevated liver function enzymes possibly related to testosterone replacement therapy

LIMITATIONS AND CAVEATS:
Compared to similar trials our trial was relatively small. Although there was statistical and clinical changes associated with testosterone replacement therapy, the translation of these findings with regard to functional gain was not addressed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No